CLINICAL TRIAL: NCT00524758
Title: Comprative Study of the Safety and Effectiveness Between Oculusgen (Ologen) Collagen Matrix Implant and Mitomycin-C in Glaucoma Filtering Surgery
Brief Title: Oculusgen (Ologen) Glaucoma MMC Control in Estonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pro Top & Mediking Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: oculusgen 2006-02-20
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Open Angle Glaucoma; Angle Closure Glaucoma; Uveitis Glaucoma; Young Age Glaucoma; Neovascular Glaucoma; High Risk Patient
Keywords: ologen; oculusgen; collagen matrix; trabeculectomy; filtering surgery; mitomycin-C; MMC; Aeon Astron
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma, Angle-Closure; Glaucoma, Neovascular | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ologen in Trabeculectomy (Experimental): Ologen in Trabeculectomy
  Interventions: Device: ologen (oculusgen) collagen matrix
- MMC in Trabeculectomy (Active Comparator): MMC in Trabeculectomy
  Interventions: Drug: MMC in Trabeculectomy

INTERVENTIONS:
Device: ologen (oculusgen) collagen matrix — Implant ologen collagen matrix on the top of sclera flap after loose stiched the sclera flap. The traditional trabeculectomy is performed.
  Other Names: ologen collagen matrix; oculusgen collagen matrix
  Arms: Ologen in Trabeculectomy
Drug: MMC in Trabeculectomy — MMC in Trabeculectomy
  Arms: MMC in Trabeculectomy

SUMMARY:
To compare the safety and effectiveness between ologen collagen matrix and mitomycin-C (MMC) in glaucoma surgery.

The ologen collagen matrix implantation procedure is same as traditional trabeculectomy except implant the ologen collagen matrix on the top of sclera flap after one loose stich the sclera flap. The MMC application is as the standard.

DETAILED DESCRIPTION:
Ologen collagen matrix is implanted on the top of sclera flap after the loose stich sclera flap is done for the filtering surgery. The concept of ologen collagen matrix is to creat the subconjunctiva bleb and modulate the wound healing for the surgery. By implanting ologen collagen matrix in the place, subconjuctival and trabdoor scars might be prevented. This is because the ologen collagen matrix is a 3-D scaffold porous structure that can guide fibroblast to grow randomly, instead of linear alignment. This can reduce the scar formation.

Doctors apply MMC for the glaucoma surgery is also trying to inhibite the scar formation. But MMC has been long time used and glaucoma specialists have not found anything to replace it.

Ologen collagen matrix concept is not INHIBITION, it is guiding and creating a physiological tissue. The successful of ologen collagen matrix may be on par with MMC but the safety and side effects will be much less.

ELIGIBILITY:
Inclusion Criteria:

* Max anti glaucoma medication failed,

Exclusion Criteria:

* Age less than 18, woman in pregnant, hemodialysis patient

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
IOP <21mmHg without anti glaucoma medication | 180 days

SECONDARY OUTCOMES:
IOP<21mmHg or IOP drops more than 30% with anti glaucoma medication | 180-day

CONTACTS AND LOCATIONS:
Overall Officials: Kuldar Kaljurand, MD, Principal Investigator — University of Tartu
Locations (1):
- Tartu University Clinics, Tartu, Estonia

REFERENCES:
- [Derived] Park J, Rittiphairoj T, Wang X, E JY, Bicket AK. Device-modified trabeculectomy for glaucoma. Cochrane Database Syst Rev. 2023 Mar 13;3(3):CD010472. doi: 10.1002/14651858.CD010472.pub3. PMID 36912740